CLINICAL TRIAL: NCT02607748
Title: 18F-fluoride (18F-NaF) Positron Emission Tomography (PET) for Identification of Ruptured and High-Risk Coronary Atherosclerotic Plaques
Brief Title: 18F-fluoride (18F-NaF) PET for Identifying Coronary Atherosclerotic Plaques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Daniel S. Berman, Chief, Nuclear Cardiology and Cardiac Imaging, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 39453
Record Dates: First submitted 2015-11-11; First posted 2015-11-18 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease; Atherosclerotic Plaque
Keywords: 18F-NaF PET; 18F-sodium fluoride PET; Coronary CTA
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic | interventions — Sodium Fluoride; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-NaF PET and coronary CTA imaging (Experimental): 18F-NaF PET and coronary CTA imaging
  Interventions: Other: 18F-NaF PET and coronary CTA imaging

INTERVENTIONS:
Other: 18F-NaF PET and coronary CTA imaging
  Other Names: 18F-NaF (sodium fluoride) PET; sodium fluoride PET; coronary CTA; CCTA; coronary CT Angiography; non-invasive coronary CT Angiography; non-invasive coronary plaque imaging

SUMMARY:
The purpose of this study is to evaluate whether 18F-NaF (sodium fluoride) Positron Emission Tomography (PET) scans can be used to identify ruptured and high-risk plaque as compared to non-invasive coronary Computed Tomography Angiography (CTA) scans and high-definition intravascular ultrasound (IVUS).

In subsets of patients, 18F-NaF PET scans and CCTA will be repeated to assess scan-rescan reproducibility.

DETAILED DESCRIPTION:
This research involves having cardiac 18F-NaF PET imaging of the heart and coronary Computed Tomographic Angiography (CTA) in a one-day visit. Three groups of patients will be enrolled: patients with Acute Coronary Syndrome, patients with stable ischemic heart disease, and asymptomatic patients with suspected coronary artery disease.

Prior to 18F-NaF administration, participants will have blood drawn to measure serum creatinine and other biomarkers related to heart disease.

All participants will undergo a 18F-NaF PET scan and a coronary CTA (which includes contrast administration). If medically appropriate, participants will have oral or intravenous beta-blocker (metoprolol) and nitroglycerin prior to CTA imaging.

Up to 10 patients will be asked to return for repeat18F-NaF PET and coronary CTA imaging 2 to 21 days after the initial scan. Up to 20 patients will be asked to return for repeat 18F-NaF PET scan and coronary CTA imaging about 6 months after the initial scan. Researchers will compare the repeat images to the initial studies.

ELIGIBILITY:
Inclusion Criteria:

Three groups of patients will be recruited for this study.

1. Acute Coronary Syndrome group: 40 patients with type 1 myocardial infarction within 21 days prior to the imaging visit and invasive coronary angiography with angiographic evidence of at least a 50% stenosis in one or more coronary arteries. Only patients undergoing PCI will be included in the study.
2. Stable Ischemic Heart Disease group: 40 patients who have undergone invasive coronary angiography within 21 days prior to the imaging visit, with history of typical angina prior to the angiogram, but no prior myocardial infarction or coronary revascularization.
3. Asymptomatic CAD group: 40 patients who have undergone Coronary Artery Calcium scanning within 6 months prior to the imaging visit, matched to the ACS patients for age, gender, and CAC score.

   * Patients in the asymptomatic CAD group must

     * have no prior CAD associated event (no prior myocardial infarction, acute coronary syndrome, coronary angiogram, or PCI),
     * have CAC between 10 to <1000, and
     * match to patients in the ACS group by gender, age by decile, and CAC category (using CAC categories of 10 to <100, 100 to <400, 400 to <1000).

Exclusion Criteria:

* Age < 18 years
* Creatinine > 1.5 mg/dL
* History of severe allergy to Iodine contrast agents
* Pregnancy
* Active atrial fibrillation
* Multiple premature ventricular or atrial contractions
* Ejection fraction <35%
* Class III congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
target-to-background ratio (TBR) uptake of 18F-NaF | one day
  a comparison of the uptake of 18F-NaF in an atherosclerotic plaque lesion compared to the background (superior vena cava)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S. Berman, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States